CLINICAL TRIAL: NCT03327181
Title: Short-chain Fatty Acid Metabolism in Chronic Obstructive Pulmonary Disease
Brief Title: Short Chain Fatty Acid Metabolism in COPD
Acronym: SCFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-0112
Record Dates: First submitted 2017-10-10; First posted 2017-10-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: short chain fatty acid metabolism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Experimental): The subject will arrive fasted. A catheter will be inserted in the arm for stable tracer SCFA infusion and blood sampling. The hand of the arm used for blood sampling will be placed in a thermostatically controlled warmed box that heats the air. Immediately after a baseline blood sample is taken, an infusion with stable tracers will be administered by the research nurse. Stable tracers are given to measure SCFA metabolism. Blood samples will be collected before and/or after infusion. Subjects will be asked to complete a list of questions regarding quality of life, mood and depression, diet, and a variety of functional measurements.
  Interventions: Dietary Supplement: short chain fatty acid tracers
- Healthy older adults (Active Comparator): The subject will arrive fasted. A catheter will be inserted in the arm for stable tracer SCFA infusion and blood sampling. The hand of the arm used for blood sampling will be placed in a thermostatically controlled warmed box that heats the air. Immediately after a baseline blood sample is taken, an infusion with stable tracers will be administered by the research nurse. Stable tracers are given to measure SCFA metabolism. Blood samples will be collected before and/or after infusion. Subjects will be asked to complete a list of questions regarding quality of life, mood and depression, diet, and a variety of functional measurements.
  Interventions: Dietary Supplement: short chain fatty acid tracers

INTERVENTIONS:
Dietary Supplement: short chain fatty acid tracers — stable tracer infusion of acetate, propionate, and butyrate

SUMMARY:
The short chain fatty acid (SCFA) metabolism has not been studied in subjects suffering from COPD. The purpose of this study is to compare the SCFA metabolism in COPD patients to healthy matched controls. This protocol is an extension of recent studies about protein digestion and absorption abnormalities in COPD patients. The investigators hypothesize that SCFA production might be lower in COPD patients than in healthy subjects.

DETAILED DESCRIPTION:
Short-chain fatty acids (SCFAs) are straight or branched-chain fatty acids produced by the intestinal microbiota mainly through fermentation of undigested carbohydrates, but also through degradation of dietary and endogenous proteins. With a share of 90 to 95 %, acetate (C2), propionate (C3), and butyrate (C4) are the most common SCFAs in the colon (3). The molar ratios of acetate to propionate to butyrate are on average approximately 60:20:20 throughout the whole colon. Several human studies tried to determine the in situ production of SCFAs by measuring their content in feces (5-8). But fecal SCFA concentrations do not accurately represent the concentrations in more proximal regions of the colon, because colonocytes absorb more than 95 % of SCFAs to use them as an energy source. Further, the measurement of plasma SCFA concentrations is inaccurate because SCFA plasma levels are low due to high metabolism in colonocytes and liver. Thus, stable isotope studies are needed to examine the colonic production and metabolic fate of SCFAs in healthy and diseased subjects.

SCFAs seem to have anti-inflammatory and immune modulating effects. In COPD an enhanced pulmonary inflammatory response causes a combination of small airways disease (e.g., obstructive bronchiolitis) and/or a destruction of lung parenchyma (emphysema). This leads to a progressive and persistent airflow limitation. Smoking and the exposure to polluted air are main risk factors causing COPD. In a mouse model, a diet rich in whey proteins attenuated emphysema through the suppression of respiratory inflammation. This might have been related to a high colonic SCFA concentration due to the diet. Young et al. proposed that in smokers SCFAs might mitigate both the innate-mediated systemic inflammation controlled by the liver and the inflammatory responses in the lung.

Moreover, Nielsen et al. found that gastrointestinal diseases are significantly more prevalent in COPD patients (15 %) than in patients with other diseases (9%). This might have an influence on the SCFA production in the colon. Gastrointestinal problems may also be assessed through the usage of validated questionnaires.

ELIGIBILITY:
Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years - 100 years
* Ability to lie in supine or elevated position for 1.5 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Inclusion criteria control subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years - 100 years
* Ability to lay in supine or elevated position for 1.5 hours
* No diagnosis of COPD
* Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Subjects 86 years and older that fail to get physician eligibility confirmation
* Insulin dependent diabetes mellitus
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day
* Use of short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

When during the period from enrollment to the test day any condition causing the subject to not meet inclusion criteria or to meet exclusion criteria, the subject will be excluded from the study.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
whole body short-chain fatty acid metabolism | -10, 2, 4, 6, 8, 10, 15, 20, 25, 30, 40, 50, 60 min
  change in whole body scfa metabolism

SECONDARY OUTCOMES:
Fat free mass measured using dual-energy x-ray absorptiometry | 1 day
  Difference in muscle mass between COPD patients and healthy older adults
Fat mass measured using dual-energy x-ray absorptiometry | 1 day
  Difference in fat mass between COPD patients and healthy older adults
Bone density measured using dual-energy x-ray absorptiometry | 1 day
  Difference in bone density between COPD patients and healthy older adults
handgrip strength dynamometry | 1 day
  Difference in handgrip strength between COPD patients and healthy older adults
Micro-respiratory pressure meter measurement | 1 day
  Difference in maximum inspiratory and expiratory pressure between COPD patients and healthy older adults
moving balance platform measurement | 1 day
  Changes in ability to maintain balance after perturbation of moving platform between COPD patients and healthy older adults. The maximum platform displacement the participant could withstand without stepping will be determined.
Group differences in attention and executive functions as measured by Trail Making Test (TMT), | 1 day
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT), | 1 day
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in somatosensory functions as measured by vibrotactile behavioral battery | 1 day
  The vibrotactile behavioral battery consists of a non-invasive set of brief tasks targeting sensory processes and inhibition. It can be used to detect neurobiological abnormalities in sensory processing. The battery of vibrotactile tasks involves the use of a small device that is designed to administer calibrated vibratory stimuli to the glabrous skin of digits 3 and 4 of the left hand and is connected to a laptop computer.
Group differences in gut function as reported by "The Gastrointestinal Symptom Rating Scale" | 1 day
  self-administered questionnaire regarding gut function and associated symptoms
Group differences in physical activity as reported by "International Physical Activity Questionnaire" | 1 day
  self-administered questionnaire regarding physical activity
COPD Assessment Test | 1 day
  self-administered questionnaire regarding impact of COPD on daily life

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951